CLINICAL TRIAL: NCT00612963
Title: Novel Rinse to Treat Oral Candidiasis in Cancer Patients "Evaluate Iocide Oral Rinse in Any Patient With Thrush, Including But Not Limited to Patients Currently Receiving or Post Radiation Therapy for Head and Neck Cancer or Patients Positive for HIV/AIDS or Transplant Patients"
Brief Title: Novel Rinse to Treat in Oral Candidiasis in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Biomedical Development Corporation (Industry)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); University of Texas (Other)
Responsible Party: Spencer Redding, DDS, Med., UTHSCSA
Other Study IDs: HSC20070023H; 5R44DE017301-03 (NIH)
Record Dates: First submitted 2008-01-30; First posted 2008-02-12 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2009-08

CONDITIONS: Candidiasis, Oral; Thrush; Candidiasis
Keywords: Candidiasis, Oral; Thrush; Candidiasis
MeSH Terms: conditions — Candidiasis, Oral; Candidiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Frio Oral Rinse — Prescription Mouth Rinse

SUMMARY:
The purpose of the study is to evaluate the efficacy of Iocide oral rinse as a treatment for Oral Candidiasis in any patient including but not limited to patients receiving radiation therapy or who have previously received radiation therapy for head and neck cancer, or patients positive for HIV/AIDS or are transplant patients.

DETAILED DESCRIPTION:
A four-week study has been designed as an assessment of the clinical cure and mycological eradication of oral Candida isolates in 40 cancer patients referred by radiation oncologists during the course of his/her treatment. An estimated 35 patients will be evaluable at the end of the study. Candida infection is defined as positive clinical signs (white plaques) with positive potassium hydroxide (KOH) preparation and positive cultures. Colonization is defined as a positive culture without signs of clinical infection.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females currently receiving or post radiation therapy for head and neck cancer;
* 18 years of age;
* With signs and symptoms of oral candidiasis as determined by investigator(s);
* Females using an effective contraception method during study.
* Patients must be able and willing to comply with study requirements, and have full understanding of all elements of, and signature and dating of, informed consent prior to initiation of protocol specified procedures.
* Participating female subjects must agree to use adequate contraceptive measures during the trial. Before entering the study, women of childbearing age will be tested for pregnancy with a urine pregnancy test.

Exclusion Criteria:

* History, or current evidence, of any significant acute or chronic medical or psychiatric condition that would render examination difficult or invalid or prevent the subject from active study participation;
* Inability to use an oral rinse;
* Use of concomitant medication that, in the opinion of the Study Director, might interfere with the outcome of the study (e.g. anabolic steroids or excessive corticosteroids, large doses of aspirin (no more than one 325 mg tablet per day), phenytoin, lithium, coumadin or Iodine containing preparations [use of iodized table salt is acceptable]). Steroids, therapeutic doses of non-steroidal anti-inflammatory agents, estrogen therapy agents and oral contraceptives are OK to use as long as the baseline dose remains steady through the end of the study;
* Use of antifungal medication in the last 30 days, purported sensitivity or allergy to iodine;
* Pregnant or nursing patients as the effect of Iocide in the fetus or infant are not established;
* History thyroid disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female volunteers who are currently receiving or post radiation therapy for head and neck cancer and currently having signs and/or symptoms of oral candidiasis
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2007-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary analysis will be "intention to treat." | 2 Weeks

SECONDARY OUTCOMES:
Clinical cure, absence of white plaque | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Spencer W. Redding, DDS, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - University of Missouri at Kansas City, School of Dentistry, Kansas City, Missouri
  - Cancer Therapy and Researh Center, San Antonio, Texas